CLINICAL TRIAL: NCT02111122
Title: A Phase II, Prospective, Randomized, Double-blind, Crossover Placebo-controlled Study of the Symptomatic Effects of Nocturnal Sodium Oxybate in Parkinson's Disease
Brief Title: Study of the Symptomatic Effects of Nocturnal Sodium Oxybate in Parkinson's Disease
Acronym: PD-Xyrem
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Christian Baumann (Other)
Responsible Party: Sponsor-Investigator, Christian Baumann, Professor dr. med., University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KEK-ZH-Nr. 2013-0239
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Sleep-wake Disturbances in Motor-phase Parkinson's Disease
Keywords: excessive daytime sleepiness; Parkinson's Disease; sleep-wake disturbances; Sodium Oxybate
MeSH Terms: conditions — Disorders of Excessive Somnolence; Parkinson Disease | interventions — Sodium Oxybate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium Oxybate (Experimental): Treatment (500mg Natrii oxybas/ml) will be administered every day at night time for 6 weeks each orally by the patient itself. If necessary, the investigator will make sure that a relative or caregiver is able to assist in daily treatment administration. The dosage starts at 3g per night and is adapted in steps of 1.5g during visits and telephone screenings and always noted in the "medication log-book". The maximal dosage is 9g per night.
  Interventions: Drug: Sodium Oxybate
- Placebo (Placebo Comparator): Treatment will be administered every day at night time for 6 weeks each orally by the patient itself. If necessary, the investigator will make sure that a relative or caregiver is able to assist in daily treatment administration. As with the active compound, placebo will be given with a starting dose of 3g per night and is adapted in steps of 1.5g during visits and telephone screenings and always noted in the "medication log-book". The maximal dosage is 9g per night.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium Oxybate
  Other Names: Brand name: Xyrem
  Arms: Sodium Oxybate
Drug: Placebo
  Arms: Placebo

SUMMARY:
Sleep wake disturbance is a common problem in Parkinson's disease patients and so far the therapeutic possibilities for symptomatic relief are limited. Small, open-label studies indicate that the use of Xyrem (gamma-hydroxybutyrate) might be of benefit in this situation.

This study is intended to show a beneficial effect of the study medication in a randomized cross-over trial, that fulfills strict scientific criteria.

DETAILED DESCRIPTION:
Background and Rationale

Non-motor symptoms as excessive daytime sleepiness (EDS) are markedly impairing quality of life in Parkinson's Disease (PD) patients. Beside the disturbing character of these symptoms, EDS for example is also linked to a decrease in cognitive abilities or mood, i.e. depression [1,2]. The most prominent cause for EDS is a disruption of nocturnal sleep [3]. Furthermore disrupted nocturnal sleep is also likely influencing quality of life of partners or caregivers. This aspect of non-motor symptoms has not been investigated in detail so far. In conclusion, we are firmly convinced that the improvement of nocturnal sleep in PD patients is a promising potential strategy to reduce several symptoms and adverse events in PD patients and their partners or caregivers. Moreover, sleep modulation is a recently introduced approach of potential neuroprotective strategies, e.g. since sleep deprivation was linked with neurodegenerative processes in the brain [4,5].

It has already been shown in a recent study that the nocturnal application of sodium oxybate in PD patients is not only improving nocturnal sleep quality, but is accompanied by a reduction in EDS [6]. There were, however, significant methodological limitations to this study, since it was a single-arm, open-label, uncontrolled study.

In summary, the nocturnal application of sodium oxybate seems to be a promising treatment for PD patients, but methodologically correct evidence is still lacking.

Investigational Product

The investigational product used in this study is Xyrem, which was approved by Swissmedic in June 2006 for the treatment of cataplexies in patients with narcolepsy. Xyrem belongs to the class of sedatives. The chemical name for sodium oxybate is sodium 4-hydroxybutyrate and its molecular formula is C4H7NaO3. Xyrem oral solution contains 500 mg of sodium oxybate per milliliter of USP Purified Water, neutralized to pH 7.5 with malic acid. It has to be taken orally at night in a split dose regime. It is eliminated mainly by metabolism with a half-life of 0.5 to 1 hour. Pharmacokinetics are nonlinear with blood levels increasing 3.8-fold as dose is doubled from 4.5 to 9 g. The pharmacokinetics are not altered with repeat dosing.

The exact mechanism of Xyrem is unknown. However, Xyrem is enhancing deep sleep and therefore strengthening nocturnal sleep. Since disturbed nocturnal sleep and EDS are major non-motor symptoms in patients suffering from PD we aim to investigate the profit of Xyrem application for PD patients (for detailed information see Arzneimittel-Kompendium der Schweiz 2012).

Clinical Data to Date

An uncontrolled open-label study administered nocturnal sodium oxybate for excessive daytime sleepiness in PD [6]. No other tested treatment so far - be it stimulants, be it continuous dopaminergic stimulation overnight - has yielded such a dramatic improvement of EDS: mean Epworth sleepiness scale values dropped down from 15.6 points (severe sleepiness, comparable to patients with narcolepsy) to 9.0 (normal values) (Table 1). In addition, sleep quality and fatigue improved as well.

In terms of safety, the Apnea-Hypopnea-Index (AHI) went up from 7 to 13, but oxygen saturations remained stable on sodium oxybate [6]. There were, however, significant methodological limitations to this study. First, it was open-label, and second, excessive daytime sleepiness was assessed only by subjective measures, i.e. with validated questionnaires.

Dose Rationale

The standard maximal dose, corresponding to the maximal dose used in this study, is 9g (corresponds to 18ml) per night in a split dose regime. As Xyrem is approved for long-term use and is only applied over 6 weeks in the current study, no specific precautions concerning the duration of intake has to be done.

The exclusion criteria in the present study meet the contraindications in case of Xyrem application listed by Swissmedic: subjects are not included in case of pregnancy, application of other CNS sedative drugs (opioids, barbiturates), severe medical conditions as liver failure, renal insufficiency, congestive heart failure and severe depression.

As most drugs, Xyrem can potentially and in few cases lead to several adverse events. Since the maximal dose is also accompanied by a higher occurrence of adverse events, the initial dose is set at 3g per night, which is even below the suggested starting dose according to the "Arzneimittelcompendium" and is carefully and stepwise increased to the individual optimal dose carefully. The key feature of a safe application is accurate monitoring of the patients, which is warranted with regular visits and phone calls in the present study.

Xyrem has been associated with potential breathing depression. In the study of Ondo et al. [6] total apneas mildly increased after the application of nocturnal sodium oxybate, whereas oxygen de-/saturation values remained stable. Nevertheless, subjects with elevated AHI or low oxygen saturation are not included in the present study (see exclusion criteria section 7.2). However, AHI will be measured before and after drug application in all subjects, allowing a better evaluation of this aspect in the future.

Up to date, there is no approved medication for sleep disturbances or EDS in PD. So far, the application of nocturnal sodium oxybate has revealed the largest improvements in PD patients. Modafinil or Rivotril have been demonstrated to have some benefits on EDS or sleep in PD patients. However, these medications are not really an alternative treatment since the effects are only moderate and the experience of their application in PD patients is still insufficient.

Risk/Benefits and Ethical Considerations

Xyrem is a drug licensed by the FDA and Swissmedic for the use in patients with narcolepsy, and its tolerability in clinical practice is very good. It is known that the use of Xyrem leads to an improvement of the quality of nocturnal sleep in patients suffering from narcolepsy, reducing EDS. In dealing with patients it is well known that sleep disturbances of any kind (endogenous as well as exogenous) impair daytime vigilance and at the same time quality of life. It is known that non-motor symptoms of PD, i.e. EDS, have a major impact on the quality of life of patients - as well as their carers. Improving nocturnal sleep would therefore be a promising possibility to enhance the patients' daytime wellbeing.

In addition to the mentioned symptomatic effect on EDS, sleep modulation might in the future emerge as a potential disease modulating strategy. Experimental animal data have shown an aggravation of neurodegenerative disease with sleep restriction (6) - it is currently under investigation if sleep modulation can work the opposite way as well.

Thereby the controlled risk of the mentioned adverse events in section 4.5 must be seen in relation to the potential benefit of improved quality of life of patients and carers as well as its potential influence on motor and non-motor symptoms and long-term disease modification.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe Parkinson's disease (Hoehn and Yahr II/III) diagnosis according to international criteria [14],
* History of disturbed nocturnal sleep and presence of EDS (ESS >10 points),
* Doses of dopaminergic and other PD treatment must have been stable for at least 14 days prior to the screening visit,
* Negative pregnancy test prior to inclusion (except in women who are surgically sterilized/hysterectomized or post-menopausal for longer than 2 years),
* Patients are capable of giving informed consent,
* Signed Informed Consent after being informed.

Exclusion Criteria:

Atypical Parkinson disorder, Parkinson's disease without response to levodopa,

* AHI >15 or oxygen saturation consistently below 90% on baseline polysomnography
* diagnosis of sleep apnoea-syndrome or COPD
* Severe dementia (MoCA<22),
* Moderate to severe depression (HADS>15).
* Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product,
* Regular use of CNS depressant substances (opioids, barbiturates) as well as melatonin and other sleep-inducing substances,
* Other clinically significant concomitant disease states (e.g., renal insufficiency (creatinin > 120 resp. GFR <40ml/min), hepatic dysfunction (GPT > 100U/l), severe cardiovascular disease, etc),
* Known or suspected non-compliance, substance or alcohol abuse (i.e. > 0.5 l wine or 1 l beer per day),
* Homeless persons,
* Women who are pregnant or breast feeding,
* Intention to become pregnant during the course of the study,
* Lack of safe contraception, defined as:

Female patients of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases.

Please note that female patients who are surgically sterilized/hysterectomized or post-menopausal for longer than 2 years are not considered as being of child bearing potential.

* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, etc. of the patient,
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons,

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Objective excessive daytime sleepiness | after 6 weeks of treatment
  mean latencies in the MSLT (multiple sleep latency test)
effect on night-time breathing | after 6 weeks of treatment
  AHI (apnoea/hypopnoea) score on polysomnography

SECONDARY OUTCOMES:
Motor function | after 6 weeks of treatment
  Part III of the Unified Parkinson's Disease Rating Scale (UPDRS) will be used to assess motor functions in PD in ON & OFF state
Subjective quality of nocturnal sleep | after 6 weeks of treatment
  assessed by the Parkinson's Disease Sleep Scale (PDSS-2) and the REM Sleep Behavior Disorder Screening Questionnaire (RBDSQ) in German. Additional questions about the change in symptoms are added to the RBDSQ and PDSS-2
Objective quality of nocturnal sleep including breathing indices | after 6 weeks of treatment
  assessed by overnight Polysomnography (PSG; using the recording system Embla N7000/M-Drive) which includes video monitoring for scoring purposes including eye movements, heart rate, muscle tone, limb movements, nasal airflow, blood oxygen saturation, breathing pattern
Overall quality of life | after 6 weeks of treatment
  The Parkinson's Disease Questionnaire (PDQ-39) in German will be used to assess changes in quality of life in PD patients
Mood | after 6 weeks of treatment
  The Parkinson's Disease Questionnaire (PDQ-39) in German will be used to assess quality of life in PD patients
Cognition | after 6 weeks of treatment
  The Montreal Cognitive Assessment (MoCA) in German will be used to quantify cognitive function by a fast and established questionnaire which is recommended by the Parkinson Study Group for use in clinical trials
Impulse control | after 6 weeks of treatment
  Impulse control and potential impulsive-compulsive disorders will be assessed by the Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease-Rating Scale (QUIP-RS) in German
Vigilance | after 6 weeks of treatment
  Vigilance will be assessed by two self-reported questionnaires by the patients, the Epworth Sleepiness Scale (ESS) and the Fatigue Severity Scale (FSS; see appendix). During the MSLT, we will perform the Sustained Attention to Response Test (SART) and the Psychomotor Vigilance Test (PVT) after the first and the third nap.
Subjective Daytime sleepiness | after 6 weeks of treatment
  In addition to the objective EDS measured by the MSLT, subjective sleepiness will be assessed prior to each nap in the course of the MSLT by the Karolinska Sleepiness Scale and the Stanford Sleepiness Scale
Sleep wake rhythm | after 6 weeks of treatment
  Sleep and physical activity levels will be recorded over 14 days by wrist actigraphy (on the non-dominant wrist; light sensor data included, Actiwatch, Respironics) [11]. We will assess the amount of activity, the amount of rest and estimate the number of naps. The recording is starting 14 days before each start of drug administration and 14 days before the end of the respective administration.
Quality of life for caregivers | after 6 weeks of treatment
  Quality of life of partners or caregivers will be assessed by the Zarit Burden of caregiver Interview (ZBCI), which is validated in its german version [12] and for Parkinson patients [13]

CONTACTS AND LOCATIONS:
Overall Officials: Christian R Baumann, MD, Principal Investigator — University of Zurich
Locations (1):
- Department of Neurology, Zurich, Switzerland

REFERENCES:
- [Derived] Buchele F, Hackius M, Schreglmann SR, Omlor W, Werth E, Maric A, Imbach LL, Hagele-Link S, Waldvogel D, Baumann CR. Sodium Oxybate for Excessive Daytime Sleepiness and Sleep Disturbance in Parkinson Disease: A Randomized Clinical Trial. JAMA Neurol. 2018 Jan 1;75(1):114-118. doi: 10.1001/jamaneurol.2017.3171. PMID 29114733